CLINICAL TRIAL: NCT00775437
Title: Compassionate Use Study of Adalimumab in Children 2 to < 4 Years Old or Age 4 and Above Weighing Less Than 15 kg With Active Juvenile Idiopathic Arthritis (JIA)
Brief Title: Active Juvenile Idiopathic Arthritis (JIA) Compassionate Use
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-444; 2009-013091-40 (EudraCT Number)
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-12

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: juvenile idiopathic arthritis; compassionate use; open label
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab (Experimental): Adalimumab 24 mg/m^2 body surface area (BSA) up to a total dose of 20 mg administered every other week (eow) by parent or designee as a single dose via subcutaneous injection at approximately the same time of day, for a minimum of 24 weeks. Participants could continue in the study until age 4 and 15 kg (US and Puerto Rico) or for up to 1 additional year after reaching age 4 and 15 kg (EU). Visits beyond Week 24 occurred every 12 weeks for those participants who continued in the study.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Adalimumab solution for injection for subcutaneous use.
  Other Names: Humira; ABT-D2E7

SUMMARY:
The main objective of this study is to evaluate the safety of adalimumab in patients 2 to < 4 years of age or ≥ 4 years of age weighing < 15 kg, with moderately to severely active polyarticular juvenile idiopathic arthritis (JIA) or polyarticular course JIA.

ELIGIBILITY:
Inclusion Criteria:

1. A parent or guardian has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), after the nature of the study has been explained and the subject's parent or legal guardian has had the opportunity to ask questions. The informed consent must be signed before any study-specific procedures are performed or before any medication is discontinued for the purpose of this study. The parent must also be willing to comply with all the requirements of this study protocol.
2. Subject has a disease diagnosis of moderately to severely active polyarticular or polyarticular course juvenile idiopathic arthritis (JIA; defined as arthritis affecting > = 5 joints at the time of treatment initiation). This corresponds to the International League of Associations for Rheumatology categories of polyarticular rheumatoid factor positive (RF+), polyarticular Rheumatoid factor negative (RF-) disease, and extended oligoarthritis disease.
3. Subject must be aged 2 to < 4 years old with moderately to severely active polyarticular JIA or polyarticular course JIA or age 4 or greater weighing < 15 kg with moderately to severely active polyarticular JIA or polyarticular course JIA, per International League of Associations for Rheumatology (ILAR) criteria.
4. Subject is judged to be in generally good health as determined by the Investigator based upon the results of medical history, laboratory profile, and physical examination performed at Screening and confirmed at Baseline. This includes, but is not limited to, a normal cardiopulmonary and normal neurological exam result.
5. Parent or legal guardian must be able and willing to administer subcutaneous (SC) injections or have a qualified person available to administer SC injections.
6. Parent or legal guardian must be willing to actively supervise storage and administration of study drug and to ensure that the time of each dose is accurately recorded in the subject's diary.
7. Subject must have negative purified protein derivative (PPD) test (or equivalent) at Screening. If subject has a positive (greater than or equal to 5mm induration) PPD test result, a chest x-ray (posterior-anterior [PA] and lateral view) must be performed. If subject has a positive test (or equivalent), has had a past ulcerative reaction to PPD placement, and/or a chest x ray consistent with tuberculosis [TB] exposure, subject may not be enrolled into the study.
8. For subjects in the European Union [EU], subject must have previously failed, had an insufficient response, or have been intolerant to at least one Disease-Modifying Anti Rheumatic Drug (DMARD).

Exclusion Criteria:

1. Subject has had prior exposure to Tysabri® (natalizumab) or Raptiva® (efalizumab) or any other biologic therapy, such as Orencia® (abatacept), Kineret® (anakinra), Actemra® (tocilizumab), Rituxan® (rituximab). Any previous use of anti-tumor necrosis factor [TNF] agents, including Enbrel® (etanercept), Remicade® (infliximab), Cimzia® (certolizumab pegol), Simponi® (golimumab), and adalimumab is also prohibited.
2. Infection(s) requiring treatment with intravenous (IV) anti-infectives within 30 days prior to Baseline Visit or oral anti-infectives within 14 days prior to the Baseline Visit.
3. Subject has undergone joint surgery within the preceding two months of the Screening Visit (at joints to be assessed within the study).
4. Subject has a previous diagnosis of a condition that could cause arthritis other than polyarticular JIA.
5. Subject has a history of an allergic reaction or significant sensitivity to constituents of the study drug, adalimumab.
6. Subject has been treated with any investigational drug of chemical or biologic nature within a minimum of 30 days or 5 half lives (whichever is longer) of the drug prior to Baseline visit. Should these biologics become approved, they would continue to be excluded.
7. Subject has a poorly controlled medical condition, such as uncontrolled diabetes, unstable heart disease, recent cerebrovascular accidents, seizure disorder, and any other condition which, in the opinion of the Investigator, would put the subject at risk by participation in the study.
8. Subject has a history of clinically significant hematologic (e.g., severe anemia, leukopenia, thrombocytopenia, a clotting disorder), renal, liver disease (e.g., fibrosis, cirrhosis, hepatitis), or active gastroenteric ulcer.
9. Subject is considered by the Investigator, for any reason, to be an unsuitable candidate for the study.
10. Subject has evidence of active TB infection.
11. Subject has history of moderate to severe congestive heart failure (New York Heart Association [NYHA] class III or IV), recent cerebrovascular accident or thrombotic event and any other condition which, in the opinion of the investigator, would put the subject at risk by participation in the protocol.
12. Evidence of dysplasia or history of malignancy (including lymphoma and leukemia).
13. History of demyelinating disease (including myelitis) or neurologic symptoms suggestive of central nervous system [CNS] demyelinating disease.
14. History of invasive fungal infection (e.g., listeriosis, histoplasmosis), active viral disorders, human immunodeficiency virus (HIV) infection.
15. Positive Hepatitis B test result.
16. Chronic recurring infections or active TB.
17. Screening laboratory and other analyses show any of the following abnormal results:

    * electrocardiogram [ECG] - with clinically significant abnormalities;
    * Aspartate transaminases (AST) or alanine transaminase (ALT) > 1.75 the upper limit of the reference range;
    * Total bilirubin >=3 mg/dL;
    * Serum creatinine > 1.6 mg/dL (convert to mmol/L).
18. Evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2009-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aileen L. Pangan, MD, Study Director — AbbVie

REFERENCES:
- [Derived] Horneff G, Seyger MMB, Arikan D, Kalabic J, Anderson JK, Lazar A, Williams DA, Wang C, Tarzynski-Potempa R, Hyams JS. Safety of Adalimumab in Pediatric Patients with Polyarticular Juvenile Idiopathic Arthritis, Enthesitis-Related Arthritis, Psoriasis, and Crohn's Disease. J Pediatr. 2018 Oct;201:166-175.e3. doi: 10.1016/j.jpeds.2018.05.042. Epub 2018 Jul 25. PMID 30054164
- [Derived] Kingsbury DJ, Bader-Meunier B, Patel G, Arora V, Kalabic J, Kupper H. Safety, effectiveness, and pharmacokinetics of adalimumab in children with polyarticular juvenile idiopathic arthritis aged 2 to 4 years. Clin Rheumatol. 2014;33(10):1433-41. doi: 10.1007/s10067-014-2498-1. Epub 2014 Feb 2. PMID 24487484
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 14 investigative sites in the Czech Republic, France, Germany, and the United States.
Pre-assignment Details: Participants age 2 to < 4 years or ≥ 4 years and under 15 kg with moderately to severely active polyarticular or polyarticular-course JIA with a parent/guardian to administer injections. The screening visit occurred between Day -28 and Day 0.
Period: Overall Study
Arm/Group | Adalimumab
Started | 32
Completed | 26
Not Completed | 6
Not completed — Loss of efficacy | 2
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.04 (0.723)
Age, Customized [Number; unit: participants]
  < 4 years | 28
  ≥ 4 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. If an AE meets any of the following criteria, it is considered a serious adverse event (SAE): Results in death, is life-threatening, results in hospitalization or the prolongation of hospitalization, is a congenital anomaly or a persistent or significant disability/incapacity, or is an important medical event requiring medical or surgical intervention to prevent a serious outcome. A treatment-emergent AE (TEAE) is defined as any AE with onset or worsening reported by a participant from the time that the first dose of adalimumab is administered until 5 half-lives (70 days) have elapsed following discontinuation of adalimumab administration (total of 32.5 months).
Time Frame: TEAEs were collected from first dose of study drug until 70 days after the last dose of study drug and before start of commercial adalimumab or other biologics (32.5 months).
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
participants
  Any Treatment-emergent AE | 29
  Any Treatment-emergent SAE | 5

2. Secondary Outcome: Mean Serum Adalimumab Trough Concentrations at Week 0, Week 12, and Week 24
Description: Adalimumab concentrations in serum were determined using a validated enzyme-linked immunoadsorbent assay (ELISA) method. The lower limit of quantitation (LLOQ) for adalimumab is 3.13 ng/mL.
Time Frame: Weeks 0, 12, and 24
Population: All participants who had samples for pharmacokinetic analysis
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Adalimumab
Number analyzed (Participants) | 15
µg/mL
  Week 0 | 0 (0)
  Week 12 | 6.97 (5.69)
  Week 24 | 7.78 (5.85)

3. Secondary Outcome: Hemoglobin: Mean Change From Baseline to Each Visit
Description: Baseline is the last value prior to the first dose of study drug. Participants with non-missing baseline and at least 1 post-baseline observation are included in the analysis. n=participants with evaluable data at given time point.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 31
g/L
  Week 12 (n=29) | 6.7 (7.32)
  Week 24 (n=29) | 6.7 (9.76)
  Week 36 (n=25) | 5.5 (9.31)
  Week 48 (n=24) | 5.3 (10.68)
  Week 60 (n=21) | 6 (10.96)
  Week 72 (n=17) | 9.5 (10.65)
  Week 84 (n=16) | 10.5 (13.69)
  Week 96 (n=11) | 8.6 (9.99)
  Week 108 (n=9) | 7.7 (8.08)
  Week 120 (n=3) | 4.7 (2.89)

4. Secondary Outcome: Hematocrit: Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: Fraction
Arm/Group | Adalimumab
Number analyzed (Participants) | 31
Fraction
  Week 12 (n=29) | 0.018 (0.0206)
  Week 24 (n=29) | 0.016 (0.0289)
  Week 36 (n=25) | 0.017 (0.0292)
  Week 48 (n=24) | 0.011 (0.0288)
  Week 60 (n=21) | 0.009 (0.0275)
  Week 72 (n=17) | 0.024 (0.0264)
  Week 84 (n=16) | 0.026 (0.0366)
  Week 96 (n=11) | 0.023 (0.0319)
  Week 108 (n=9) | 0.018 (0.0273)
  Week 120 (n=3) | 0.008 (0.0082)

5. Secondary Outcome: Red Blood Cell (RBC) Count: Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: x10˄12/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 31
x10˄12/L
  Week 12 (n=29) | 0.15 (0.231)
  Week 24 (n=29) | 0.08 (0.308)
  Week 36 (n=25) | 0.098 (0.277)
  Week 48 (n=24) | 0.05 (0.213)
  Week 60 (n=21) | 0.07 (0.296)
  Week 72 (n=17) | 0.1 (0.187)
  Week 84 (n=16) | 0.06 (0.228)
  Week 96 (n=11) | 0.08 (0.343)
  Week 108 (n=9) | 0.1 (0.32)
  Week 120 (n=3) | 0.03 (0.153)

6. Secondary Outcome: Platelets: Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: x10˄9/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 31
x10˄9/L
  Week 12 (n=29) | -35 (145.44)
  Week 24 (n=29) | -57.7 (140.82)
  Week 36 (n=25) | -75.2 (148.51)
  Week 48 (n=23) | -21 (174.17)
  Week 60 (n=21) | -46.7 (125.71)
  Week 72 (n=17) | -51.1 (111.11)
  Week 84 (n=15) | -58.5 (127.29)
  Week 96 (n=11) | -49.2 (142.73)
  Week 108 (n=9) | -30.4 (137.84)
  Week 120 (n=3) | 20 (185.95)

7. Secondary Outcome: White Blood Cell (WBC) Count: Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: x10^9/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 31
x10^9/L
  Week 12 (n=29) | 0.19 (3.959)
  Week 24 (n=29) | -0.25 (3.756)
  Week 36 (n=25) | -0.42 (4.632)
  Week 48 (n=24) | 0.3 (4.804)
  Week 60 (n=21) | 0.25 (2.183)
  Week 72 (n=17) | 0.66 (3.225)
  Week 84 (n=16) | 0.18 (2.944)
  Week 96 (n=11) | 0.55 (2.757)
  Week 108 (n=9) | -0.76 (4.166)
  Week 120 (n=3) | 1.8 (3.651)

8. Secondary Outcome: Neutrophils: Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: x10˄9/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 31
x10˄9/L
  Week 12 (n=29) | -0.138 (2.9819)
  Week 24 (n=29) | -0.619 (3.0082)
  Week 36 (n=25) | -0.586 (3.7363)
  Week 48 (n=24) | 0.065 (3.4433)
  Week 60 (n=21) | 0.222 (2.0937)
  Week 72 (n=17) | -0.169 (2.6167)
  Week 84 (n=16) | -0.206 (2.0077)
  Week 96 (n=11) | 0.293 (2.511)
  Week 108 (n=9) | -0.39 (3.1702)
  Week 120 (n=3) | 2.47 (3.2658)

9. Secondary Outcome: Lymphocytes: Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: x10˄9/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 31
x10˄9/L
  Week 12 (n=29) | 0.371 (2.3523)
  Week 24 (n=29) | 0.292 (1.9345)
  Week 36 (n=25) | 0.176 (1.962)
  Week 48 (n=24) | 0.186 (1.9584)
  Week 60 (n=21) | -0.034 (1.6129)
  Week 72 (n=17) | 0.636 (1.7404)
  Week 84 (n=16) | 0.306 (1.5143)
  Week 96 (n=11) | 0.006 (1.9402)
  Week 108 (n=9) | -0.46 (2.4315)
  Week 120 (n=3) | -0.67 (1.8041)

10. Secondary Outcome: Monocytes: Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: x10^9/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 31
x10^9/L
  Week 12 (n=29) | -0.032 (0.3051)
  Week 24 (n=29) | 0.081 (0.4547)
  Week 36 (n=25) | 0.028 (0.2978)
  Week 48 (n=24) | -0.006 (0.2718)
  Week 60 (n=21) | 0.08 (0.1831)
  Week 72 (n=17) | 0.113 (0.2054)
  Week 84 (n=16) | 0.061 (0.2594)
  Week 96 (n=11) | 0.089 (0.2295)
  Week 108 (n=9) | 0.096 (0.3248)
  Week 120 (n=3) | 0.057 (0.0777)

11. Secondary Outcome: Eosinophils: Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: x10^9/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 31
x10^9/L
  Week 12 (n=29) | -0.004 (0.1771)
  Week 24 (n=29) | -0.006 (0.1545)
  Week 36 (n=25) | -0.052 (0.1374)
  Week 48 (n=24) | 0.056 (0.2773)
  Week 60 (n=21) | -0.015 (0.1363)
  Week 72 (n=17) | 0.069 (0.1886)
  Week 84 (n=16) | 0.016 (0.1631)
  Week 96 (n=11) | 0.158 (0.3207)
  Week 108 (n=9) | -0.002 (0.0864)
  Week 120 (n=3) | -0.063 (0.0929)

12. Secondary Outcome: Basophils: Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: x10^9/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 31
x10^9/L
  Week 12 (n=29) | -0.012 (0.0299)
  Week 24 (n=29) | -0.002 (0.0272)
  Week 36 (n=25) | 0.003 (0.0244)
  Week 48 (n=24) | 0.005 (0.0412)
  Week 60 (n=21) | -0.003 (0.0256)
  Week 72 (n=17) | 0.007 (0.031)
  Week 84 (n=16) | -0.001 (0.0171)
  Week 96 (n=11) | -0.003 (0.0205)
  Week 108 (n=9) | -0.001 (0.0117)
  Week 120 (n=3) | 0.003 (0.0306)

13. Secondary Outcome: Alanine Aminotransferase (SGPT/ALT): Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 30
U/L
  Week 12 (n=27) | 0.5 (9.96)
  Week 24 (n=28) | -1.1 (17.13)
  Week 36 (n=25) | 0 (29.82)
  Week 48 (n=24) | -4.5 (24.81)
  Week 60 (n=21) | -2 (10.25)
  Week 72 (n=16) | -1.8 (10.1)
  Week 84 (n=16) | -0.5 (14.56)
  Week 96 (n=11) | -3.9 (15.4)
  Week 108 (n=9) | -2.4 (6.31)
  Week 120 (n=3) | -14.3 (23.12)

14. Secondary Outcome: Aspartate Aminotransferase (SGOT/AST): Mean Change From Baseline to Each Visit
Description: Baseline is the last value prior to the first dose of study drug.Participants with non-missing baseline and at least 1 post-baseline observation are included in the analysis. n=participants with evaluable data at given time point.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 30
U/L
  Week 12 (n=26) | 2.8 (7.56)
  Week 24 (n=28) | -0.6 (8.82)
  Week 36 (n=25) | 2 (23.26)
  Week 48 (n=24) | -0.7 (16.13)
  Week 60 (n=21) | -0.4 (7.63)
  Week 72 (n=16) | 0.3 (7.36)
  Week 84 (n=16) | -0.4 (6.89)
  Week 96 (n=10) | 1.5 (11.48)
  Week 108 (n=9) | 0.4 (6.21)
  Week 120 (n=3) | -8.3 (11.93)

15. Secondary Outcome: Alkaline Phosphatase (ALP): Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 30
U/L
  Week 12 (n=27) | 15.7 (64.65)
  Week 24 (n=28) | 10.6 (68.75)
  Week 36 (n=25) | 23.2 (73.28)
  Week 48 (n=24) | 21.7 (73.03)
  Week 60 (n=21) | 17.9 (85.55)
  Week 72 (n=16) | 17.9 (83.52)
  Week 84 (n=16) | 31.5 (89.3)
  Week 96 (n=11) | 59.4 (57.65)
  Week 108 (n=9) | -6.3 (100.72)
  Week 120 (n=3) | -72.3 (169.19)

16. Secondary Outcome: Creatine Phosphokinase: Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 30
U/L
  Week 12 (n=27) | 17.2 (50.48)
  Week 24 (n=27) | 7 (30.79)
  Week 36 (n=25) | 24.8 (44.5)
  Week 48 (n=24) | 18.4 (54.02)
  Week 60 (n=21) | 26.6 (65.48)
  Week 72 (n=16) | 41.6 (40.63)
  Week 84 (n=16) | 36.4 (53.64)
  Week 96 (n=11) | 28.7 (41.79)
  Week 108 (n=9) | 7.2 (22.97)
  Week 120 (n=3) | 14 (40.73)

17. Secondary Outcome: Total Bilirubin: Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 30
µmol/L
  Week 12 (n=27) | 1.2 (2.42)
  Week 24 (n=28) | 0.6 (1.59)
  Week 36 (n=25) | 0.6 (1.61)
  Week 48 (n=24) | 0.9 (2.4)
  Week 60 (n=21) | 1 (2.09)
  Week 72 (n=16) | 0.2 (1.25)
  Week 84 (n=16) | 0.5 (2.36)
  Week 96 (n=11) | 0.7 (1.62)
  Week 108 (n=9) | 1.1 (2.71)
  Week 120 (n=3) | 2.3 (0.58)

18. Secondary Outcome: Creatinine: Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 30
µmol/L
  Week 12 (n=27) | 1.7 (5.98)
  Week 24 (n=28) | 0.5 (5.3)
  Week 36 (n=25) | 0.3 (5.84)
  Week 48 (n=24) | 2.5 (7.8)
  Week 60 (n=21) | 2.8 (5.79)
  Week 72 (n=16) | 3.4 (6.96)
  Week 84 (n=16) | 4 (6.37)
  Week 96 (n=11) | 3.2 (5.53)
  Week 108 (n=9) | 6.2 (6.7)
  Week 120 (n=3) | 8.7 (5.51)

19. Secondary Outcome: Uric Acid: Mean Change From Baseline to Each Visit
Description: as for outcome 3
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 30
µmol/L
  Week 12 (n=27) | 1.7 (48.24)
  Week 24 (n=27) | 6.5 (47.93)
  Week 36 (n=25) | 2.5 (41.77)
  Week 48 (n=24) | 5.6 (45.62)
  Week 60 (n=21) | 1.9 (30.86)
  Week 72 (n=16) | -0.9 (43.53)
  Week 84 (n=16) | -4.5 (46.76)
  Week 96 (n=11) | 13.3 (36.39)
  Week 108 (n=9) | -10.1 (33.55)
  Week 120 (n=3) | -7 (27.78)

20. Secondary Outcome: Percentage of Participants Achieving Pediatric American College of Rheumatology (PedACR) 30% Response (PedACR30)
Description: The PedACR30 response is defined by the PedACR as ≥30% improvement in at least 3 of 6 JIA core set criteria, and ≥30% worsening in ≤1 of 6 JIA core set criteria. The 6 variables for the JIA core set criteria are Physician's Global Assessment (PGA) of participant's disease activity, Parent's Global Assessment of participant's disease activity, number of active joints (joints with swelling not due to deformity or joints with loss of passive motion [LOM] and joints with pain on passive motion [POM], tenderness, or both), number of joints with LOM, Disability Index of Child Health Assessment Questionnaire (DICHAQ), and C-reactive protein (CRP). Baseline is the last value prior to the first dose of study drug. Missing data were imputed up to Week 60 using last observation carried forward (LOCF) and non-responder imputation (NRI); observed values are presented for timepoints past Week 60. n=number of participants for either observed or imputed methods at given time point.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
percentage of participants
  Week 12 Observed (n=31) | 93.5
  Week 12 NRI (n=32) | 90.6
  Week 12 LOCF (n=31) | 93.5
  Week 24 Observed (n=30) | 90
  Week 24 NRI (n=32) | 84.4
  Week 24 LOCF (n=31) | 90.3
  Week 36 Observed (n=27) | 92.6
  Week 36 NRI (n=32) | 78.1
  Week 36 LOCF (n=31) | 93.5
  Week 48 Observed (n=24) | 83.3
  Week 48 NRI (n=32) | 62.5
  Week 48 LOCF (n=31) | 83.9
  Week 60 Observed (n=20) | 90
  Week 60 NRI (n=32) | 56.3
  Week 60 LOCF (n=31) | 87.1
  Week 72 Observed (n=17) | 100
  Week 84 Observed (n=17) | 100
  Week 96 Observed (n=13) | 92.3
  Week 108 Observed (n=9) | 88.9
  Week 120 Observed (n=3) | 100

21. Secondary Outcome: Percentage of Participants Achieving Pediatric American College of Rheumatology (PedACR) 50% Response (PedACR50)
Description: The PedACR50 response is defined by the PedACR as ≥ 50% improvement in at least 3 of 6 JIA core set criteria, and ≥ 30% worsening in not more than 1 of 6 JIA core set criteria. The 6 variables for the JIA core set criteria include PGA of participant's disease activity, Parent's Global Assessment of participant's disease activity, number of active joints (joints with swelling not due to deformity or joints with LOM and joints with POM, tenderness, or both), number of joints with LOM, DICHAQ, and CRP. Baseline is the last value prior to the first dose of study drug. Missing data were imputed up to Week 60 using LOCF and by NRI; observed values are presented for timepoints past Week 60. n=number of participants for either observed or imputed methods at given time point.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
percentage of participants
  Week 12 Observed (n=31) | 90.3
  Week 12 NRI (n=32) | 87.5
  Week 12 LOCF (n=31) | 90.3
  Week 24 Observed (n=30) | 83.3
  Week 24 NRI (n=32) | 78.1
  Week 24 LOCF (n=31) | 83.9
  Week 36 Observed (n=27) | 88.9
  Week 36 NRI (n=32) | 75
  Week 36 LOCF (n=31) | 90.3
  Week 48 Observed (n=24) | 79.2
  Week 48 NRI (n=32) | 59.4
  Week 48 LOCF (n=31) | 80.6
  Week 60 Observed (n=20) | 80
  Week 60 NRI (n=32) | 50
  Week 60 LOCF (n=31) | 80.6
  Week 72 Observed (n=17) | 100
  Week 84 Observed (n=17) | 94.1
  Week 96 Observed (n=13) | 92.3
  Week 108 Observed (n=9) | 88.9
  Week 120 Observed (n=3) | 100

22. Secondary Outcome: Percentage of Participants Achieving Pediatric American College of Rheumatology (PedACR) 70% Response (PedACR70)
Description: The PedACR70 response is defined by the PedACR as ≥ 70% improvement in at least 3 of 6 JIA core set criteria, and ≥ 30% worsening in not more than 1 of 6 JIA core set criteria. The 6 variables for the JIA core set criteria include PGA of participant's disease activity, Parent's Global Assessment of participant's disease activity, number of active joints (joints with swelling not due to deformity or joints with LOM and joints with POM, tenderness, or both), number of joints with LOM, DICHAQ, and CRP. Baseline is the last value prior to the first dose of study drug. Missing data were imputed up to Week 60 using LOCF and by NRI; observed values are presented for timepoints past Week 60. n=number of participants for either observed or imputed methods at given time point.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
percentage of participants
  Week 12 Observed (n=31) | 61.3
  Week 12 NRI (n=32) | 59.4
  Week 12 LOCF (n=31) | 61.3
  Week 24 Observed (n=30) | 73.3
  Week 24 NRI (n=32) | 68.8
  Week 24 LOCF (n=31) | 74.2
  Week 36 Observed (n=27) | 66.7
  Week 36 NRI (n=32) | 56.3
  Week 36 LOCF (n=31) | 67.7
  Week 48 Observed (n=24) | 75
  Week 48 NRI (n=32) | 56.3
  Week 48 LOCF (n=31) | 74.2
  Week 60 Observed (n=20) | 70
  Week 60 NRI (n=32) | 43.8
  Week 60 LOCF (n=31) | 71
  Week 72 Observed (n=17) | 76.5
  Week 84 Observed (n=17) | 82.4
  Week 96 Observed (n=13) | 76.9
  Week 108 Observed (n=9) | 77.8
  Week 120 Observed (n=3) | 100

23. Secondary Outcome: Percentage of Participants Achieving Pediatric American College of Rheumatology (PedACR) 90% Response (PedACR90)
Description: The PedACR90 response is defined by the PedACR as ≥ 90% improvement in at least 3 of 6 JIA core set criteria, and ≥ 30% worsening in not more than 1 of 6 JIA core set criteria. The 6 variables for the JIA core set criteria include PGA of participant's disease activity, Parent's Global Assessment of participant's disease activity, number of active joints (joints with swelling not due to deformity or joints with LOM and joints with POM, tenderness, or both), number of joints with LOM, DICHAQ, and CRP. Baseline is the last value prior to the first dose of study drug. Missing data were imputed up to Week 60 using LOCF and by NRI; observed values are presented for timepoints past Week 60. n=number of participants for either observed or imputed methods at given time point.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
percentage of participants
  Week 12 Observed (n=31) | 38.7
  Week 12 NRI (n=32) | 37.5
  Week 12 LOCF (n=31) | 38.7
  Week 24 Observed (n=30) | 36.7
  Week 24 NRI (n=32) | 34.4
  Week 24 LOCF (n=31) | 35.5
  Week 36 Observed (n=27) | 51.9
  Week 36 NRI (n=32) | 43.8
  Week 36 LOCF (n=31) | 51.6
  Week 48 Observed (n=24) | 62.5
  Week 48 NRI (n=32) | 46.9
  Week 48 LOCF (n=31) | 58.1
  Week 60 Observed (n=20) | 50
  Week 60 NRI (n=32) | 31.3
  Week 60 LOCF (n=31) | 51.6
  Week 72 Observed (n=17) | 64.7
  Week 84 Observed (n=17) | 64.7
  Week 96 Observed (n=13) | 61.5
  Week 108 Observed (n=9) | 66.7
  Week 120 Observed (n=3) | 100

24. Secondary Outcome: Physician's Global Assessment of Disease Activity: Mean Change From Baseline to Each Visit
Description: The physician's assessment of participant's overall disease activity on a visual analog scale (VAS). The VAS is a 100 mm scale, with scores ranging from 0 (very good) to 100 (very bad). Baseline is defined as the last nonmissing value prior to the first dose of study drug. Participants with nonmissing Baseline and at least 1 postbaseline observation are included in the analysis. n=participants with a nonmissing value at baseline and each visit.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=31) | -41.4 (21.2)
  Week 24 (n=30) | -45.3 (21.32)
  Week 36 (n=28) | -43 (23.9)
  Week 48 (n=24) | -46.5 (18.35)
  Week 60 (n=21) | -42.7 (28.17)
  Week 72 (n=17) | -51.1 (19.53)
  Week 84 (n=17) | -50.5 (16.77)
  Week 96 (n=13) | -47.5 (24.42)
  Week 108 (n=9) | -48.3 (28.24)
  Week 120 (n=3) | -56.3 (5.13)

25. Secondary Outcome: Parent's Global Assessment of Disease Activity: Mean Change From Baseline to Each Visit
Description: The parent's assessment of how the participant's arthritis is doing overall on a VAS. The VAS is a 100 mm scale, with scores ranging from 0 (very good) to 100 (very bad). Baseline is defined as the last nonmissing value prior to the first dose of study drug. Participants with nonmissing Baseline and at least 1 postbaseline observation are included in the analysis. n=participants with a nonmissing value at baseline and each visit.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=31) | -28.1 (29.91)
  Week 24 (n=30) | -32.2 (29.74)
  Week 36 (n=27) | -35.1 (27.42)
  Week 48 (n=24) | -35.6 (32.19)
  Week 60 (n=21) | -34.5 (33.31)
  Week 72 (n=17) | -43.8 (25.58)
  Week 84 (n=17) | -42.6 (28.62)
  Week 96 (n=13) | -45.8 (29.1)
  Week 108 (n=9) | -39.9 (37.54)
  Week 120 (n=3) | -47.7 (34.96)

26. Secondary Outcome: Disability Index of Child Health Assessment Questionnaire (DICHAQ): Mean Change From Baseline to Each Visit
Description: The DICHAQ is a self-reported participant-oriented outcome measure, calculated as the mean of the following 8 category scores (range: 0 to 3): Dressing and Grooming, Arising, Eating, Walking, Hygiene, Reach, Grip, and Activities. The score of each category is calculated as the maximum of the scores for the questions within that category. If aids and devices and/or help from another person are used for a category, a lower category score is adjusted to 2 for that category. A participant must have scores for at least 6 categories in order to compute the DICHAQ score. Total score is derived as average of all categories: 0 (no disability) to 3 (complete disability). Baseline is the last value prior to the first dose of study drug. Baseline is defined as the last nonmissing value prior to the first dose of study drug. Participants with nonmissing Baseline and at least 1 postbaseline observation are included in the analysis. n=participants with a nonmissing value at baseline and each visit.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=31) | -0.5 (0.64)
  Week 24 (n=30) | -0.5 (0.69)
  Week 36 (n=27) | -0.6 (0.7)
  Week 48 (n=24) | -0.6 (0.68)
  Week 60 (n=21) | -0.6 (0.71)
  Week 72 (n=16) | -0.9 (0.64)
  Week 84 (n=17) | -0.9 (0.68)
  Week 96 (n=13) | -0.8 (0.56)
  Week 108 (n=9) | -0.8 (0.63)
  Week 120 (n=3) | -0.8 (1.09)

27. Secondary Outcome: Active Joint Counts (AJC73): Mean Change From Baseline to Each Visit
Description: A joint assessment was recorded at all study visits to assess the number of active joints, with a total possible score of 0 (no active joints) to 73 (all active joints). Active joints are defined as joints with positive results for tenderness, swelling, pain on passive motion, or limitation of passive motion. Baseline is defined as the last nonmissing value prior to the first dose of study drug. Participants with nonmissing Baseline and at least 1 postbaseline observation are included in the analysis. n=participants with a nonmissing value at baseline and each visit.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 2 (n=32) | -5 (6.58)
  Week 4 (n=32) | -6.1 (6.69)
  Week 8 (n=32) | -7 (5.24)
  Week 12 (n=31) | -7.3 (4.52)
  Week 16 (n=31) | -7.1 (5.87)
  Week 20 (n=29) | -8 (5.68)
  Week 24 (n=30) | -7.2 (5.6)
  Week 36 (n=28) | -7.3 (5.21)
  Week 48 (n=24) | -8 (5.5)
  Week 60 (n=20) | -9.5 (7.5)
  Week 72 (n=17) | -10.2 (6.64)
  Week 84 (n=17) | -10.4 (7.57)
  Week 96 (n=13) | -8.9 (7.04)
  Week 108 (n=9) | -5.9 (3.33)
  Week 120 (n=3) | -7.3 (2.08)

28. Secondary Outcome: Limitation of Passive Motion (LOM69) Joint Count: Mean Change From Baseline to Each Visit
Description: Sixty-nine joints were assessed by physical examination. The joints to be examined for LOM were the same as those examined for tenderness, except that the sacroiliac, sternoclavicular, and acromio clavicular joints were excluded. LOM of the joint was classified as present ("1"), absent ("0"), or replaced/injected ("9"). Scores range from 0 to 621, with higher scores representing higher disease activity. Baseline is defined as the last nonmissing value prior to the first dose of study drug. Participants with nonmissing Baseline and at least 1 postbaseline observation are included in the analysis. n=participants with a nonmissing value at baseline and each visit.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 2 (n=32) | -4.5 (7.14)
  Week 4 (n=32) | -5.4 (6.48)
  Week 8 (n=32) | -5.3 (5.02)
  Week 12 (n=31) | -5.6 (4.8)
  Week 16 (n=31) | -6.3 (6.31)
  Week 20 (n=29) | -6.8 (6.63)
  Week 24 (n=30) | -5.6 (5.54)
  Week 36 (n=28) | -5.1 (5.29)
  Week 48 (n=24) | -5.5 (7.06)
  Week 60 (n=20) | -5.5 (8.31)
  Week 72 (n=17) | -6.9 (7.84)
  Week 84 (n=17) | -8.4 (6.9)
  Week 96 (n=13) | -7.5 (6.73)
  Week 108 (n=9) | -5.2 (3.96)
  Week 120 (n=3) | -6 (2.65)

29. Secondary Outcome: C-reactive Protein (CRP): Mean Change From Baseline to Each Visit
Description: CRP is a laboratory parameter and considered as an efficacy variable. CRP is a general marker of inflammation that is sensitive to acute changes in inflammatory response. CRP is reported using mg/dL. Baseline is defined as the last nonmissing value prior to the first dose of study drug. Participants with nonmissing Baseline and at least 1 postbaseline observation are included in the analysis. n=participants with a nonmissing value at baseline and each visit.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
mg/dL
  Week 12 (n=28) | -0.6 (2.65)
  Week 24 (n=28) | -0.2 (3.2)
  Week 36 (n=25) | -0.4 (3.08)
  Week 48 (n=23) | 0.4 (2.68)
  Week 60 (n=20) | -0.3 (1.83)
  Week 72 (n=17) | -0.7 (1.25)
  Week 84 (n=17) | -0.7 (1.47)
  Week 96 (n=12) | 0.1 (1.6)
  Week 108 (n=9) | 0.2 (1.93)
  Week 120 (n=3) | 0.3 (0.28)

30. Secondary Outcome: Tender Joint Count (TJC75): Mean Change From Baseline to Each Visit
Description: Seventy-five joints or regions were assessed by pressure and joint manipulation on physical examination. Joint tenderness was classified as either present ("1"), absent ("0") or replaced/injected ("9"). Scores range from 0 to 675, with higher scores representing higher disease activity. Baseline is defined as the last nonmissing value prior to the first dose of study drug. Participants with nonmissing Baseline and at least 1 postbaseline observation are included in the analysis. n=participants with a nonmissing value at baseline and each visit.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 2 (n=32) | -2.3 (4.62)
  Week 4 (n=32) | -2.8 (4.48)
  Week 8 (n=32) | -3.1 (4.31)
  Week 12 (n=31) | -2.7 (5.09)
  Week 16 (n=31) | -3.5 (4.77)
  Week 20 (n=29) | -3.9 (5.09)
  Week 24 (n=30) | -3 (5.54)
  Week 36 (n=28) | -2.9 (5.65)
  Week 48 (n=24) | -4.4 (4.85)
  Week 60 (n=20) | -4.5 (5.85)
  Week 72 (n=17) | -5.3 (5.53)
  Week 84 (n=17) | -4.8 (5.2)
  Week 96 (n=13) | -4 (5.46)
  Week 108 (n=9) | -1.1 (4.73)
  Week 120 (n=3) | -1.3 (2.31)

31. Secondary Outcome: Swollen Joint Count (SJC66): Mean Change From Baseline to Each Visit
Description: Sixty-six joints were assessed by physical examination. The joints to be examined for swelling were the same as those examined for tenderness, except that the hip, subtalar, sacroiliac, lumbar spine, thoracic spine, and cervical spine joints were excluded. Joint swelling was classified as present ("1"), absent ("0") or replaced/injected ("9"). Scores range from 0 to 594, with higher scores representing higher disease activity. Baseline is defined as the last nonmissing value prior to the first dose of study drug. Participants with nonmissing Baseline and at least 1 postbaseline observation are included in the analysis. n=participants with a nonmissing value at baseline and each visit.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 2 (n=32) | -4.5 (6.46)
  Week 4 (n=32) | -5.3 (6.63)
  Week 8 (n=32) | -6 (5.32)
  Week 12 (n=31) | -6.2 (4.24)
  Week 16 (n=31) | -6.1 (6.59)
  Week 20 (n=29) | -6.9 (5.62)
  Week 24 (n=30) | -6.3 (5.83)
  Week 36 (n=28) | -6.2 (4.73)
  Week 48 (n=24) | -6.7 (5.34)
  Week 60 (n=20) | -8.4 (7.15)
  Week 72 (n=17) | -8.9 (6.06)
  Week 84 (n=17) | -9.4 (7.15)
  Week 96 (n=13) | -8.5 (6.89)
  Week 108 (n=9) | -5.8 (3.31)
  Week 120 (n=3) | -7.3 (2.08)

32. Secondary Outcome: Pain on Passive Motion (POM75) Joint Count: Mean Change From Baseline to Each Visit
Description: Seventy-five joints were assessed by physical examination. The joints to be examined for POM were the same as those examined for tenderness. POM of the joint was classified as present ("1"), absent ("0"), or replaced/injected ("9"). Scores range from 0 to 675, with higher scores representing higher disease activity. Baseline is defined as the last nonmissing value prior to the first dose of study drug. Participants with nonmissing Baseline and at least 1 postbaseline observation are included in the analysis. n=participants with a nonmissing value at baseline and each visit.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 2 (n=32) | -3.3 (4.5)
  Week 4 (n=32) | -4 (4.01)
  Week 8 (n=32) | -4.6 (5.17)
  Week 12 (n=31) | -4.9 (4.59)
  Week 16 (n=31) | -4.9 (4.6)
  Week 20 (n=29) | -5.4 (4.81)
  Week 24 (n=30) | -4.1 (7.32)
  Week 36 (n=28) | -4.3 (7.34)
  Week 48 (n=24) | -5.8 (4.42)
  Week 60 (n=20) | -5.9 (5.25)
  Week 72 (n=17) | -6.4 (5.41)
  Week 84 (n=17) | -6.1 (5.34)
  Week 96 (n=13) | 5.7 (5.12)
  Week 108 (n=9) | -3.6 (5.85)
  Week 120 (n=3) | -5.3 (1.53)

33. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Global Health Category: Mean Change From Baseline to Each Visit
Description: The CHQ-PF50 is a participant-reported outcome measure that includes 50 questions related to physical and mental health, social limitations, and impact on parents and family. Scores for each category were converted to a scale from 0 (implies higher disease activity) to 100 (implies lower disease activity). Baseline is defined as the last nonmissing value prior to the first dose of study drug. Participants with nonmissing Baseline and at least 1 postbaseline observation are included in the analysis. n=participants with a nonmissing value at baseline and each visit.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=29) | 17.1 (29.48)
  Week 24 (n=28) | 24.3 (25.77)
  Week 36 (n=24) | 25 (27.27)
  Week 48 (n=22) | 30.9 (23.79)
  Week 60 (n=19) | 21.8 (27.35)
  Week 72 (n=17) | 31.5 (24.86)
  Week 84 (n=17) | 26.2 (25.89)
  Week 96 (n=11) | 32.7 (20.66)
  Week 108 (n=8) | 36.9 (19.99)
  Week 120 (n=3) | 45 (17.32)

34. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Physical Functioning Category: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=31) | 30.6 (32.14)
  Week 24 (n=30) | 31.6 (31.91)
  Week 36 (n=27) | 36.4 (31.26)
  Week 48 (n=23) | 31.5 (28.39)
  Week 60 (n=21) | 29 (32.3)
  Week 72 (n=16) | 40.6 (27)
  Week 84 (n=17) | 40 (30.44)
  Week 96 (n=13) | 34.3 (27.88)
  Week 108 (n=9) | 37 (27.92)
  Week 120 (n=3) | 53.7 (8.49)

35. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Role/Social Limitations/Emotional/Behavioral Category: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=23) | 20.8 (32.53)
  Week 24 (n=22) | 17.7 (29.43)
  Week 36 (n=20) | 17.2 (25.86)
  Week 48 (n=18) | 16 (27.28)
  Week 60 (n=16) | 20.8 (31.91)
  Week 72 (n=13) | 26.5 (32.25)
  Week 84 (n=13) | 20.5 (33.29)
  Week 96 (n=9) | 30.9 (32.76)
  Week 108 (n=7) | 23.8 (25.2)
  Week 120 (n=2) | 33.3 (47.14)

36. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Role/Social Limitations - Physical Category: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=21) | 28.6 (32.97)
  Week 24 (n=20) | 31.7 (35)
  Week 36 (n=18) | 30.6 (39.3)
  Week 48 (n=17) | 27.5 (37.24)
  Week 60 (n=15) | 34.4 (39.07)
  Week 72 (n=12) | 36.1 (41.34)
  Week 84 (n=12) | 34.7 (43.5)
  Week 96 (n=8) | 41.7 (37.8)
  Week 108 (n=6) | 47.2 (37.14)
  Week 120 (n=1) | 66.7 (0)

37. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Bodily Pain/Discomfort Category: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=30) | 35 (30.6)
  Week 24 (n=29) | 36.2 (32.99)
  Week 36 (n=26) | 38.8 (27.76)
  Week 48 (n=23) | 41.7 (29.64)
  Week 60 (n=20) | 39 (34.78)
  Week 72 (n=17) | 48.2 (20.38)
  Week 84 (n=17) | 41.2 (25.47)
  Week 96 (n=13) | 42.3 (23.51)
  Week 108 (n=9) | 41.1 (37.56)
  Week 120 (n=3) | 50 (17.32)

38. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Behavior Category: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=29) | 5.6 (15.78)
  Week 24 (n=28) | 4.2 (13.58)
  Week 36 (n=27) | 0.4 (16.87)
  Week 48 (n=24) | 3.6 (17.04)
  Week 60 (n=21) | -0.3 (13.95)
  Week 72 (n=17) | 0.1 (16.44)
  Week 84 (n=17) | 1.5 (13.97)
  Week 96 (n=13) | 7.1 (11.81)
  Week 108 (n=9) | 8.9 (10.46)
  Week 120 (n=3) | -6.1 (31.28)

39. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Global Behavior Item: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=19) | 4.5 (18.17)
  Week 24 (n=19) | 10.8 (17.66)
  Week 36 (n=18) | 9.2 (25.04)
  Week 48 (n=16) | 4.1 (18.55)
  Week 60 (n=13) | -3.5 (20.35)
  Week 72 (n=10) | 2 (15.31)
  Week 84 (n=11) | -5 (14.32)
  Week 96 (n=9) | 0 (17.68)
  Week 108 (n=6) | -4.2 (10.21)
  Week 120 (n=1) | -25 (0)

40. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Mental Health Category: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=31) | 3.5 (11.12)
  Week 24 (n=30) | 3.5 (10.76)
  Week 36 (n=27) | 4.1 (14.01)
  Week 48 (n=24) | 5.4 (11.88)
  Week 60 (n=21) | 2.1 (14.02)
  Week 72 (n=17) | 5 (12.37)
  Week 84 (n=17) | 2.6 (8.5)
  Week 96 (n=13) | 4.2 (11.88)
  Week 108 (n=9) | -0.8 (15)
  Week 120 (n=3) | -3.3 (20.21)

41. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Self Esteem Category: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=23) | 10.6 (23.91)
  Week 24 (n=22) | 10.5 (24.75)
  Week 36 (n=19) | 16.8 (22.02)
  Week 48 (n=16) | 15.2 (22.6)
  Week 60 (n=14) | 10.2 (22.53)
  Week 72 (n=13) | -2.8 (31.78)
  Week 84 (n=13) | 9.4 (18.52)
  Week 96 (n=9) | 6.9 (19.87)
  Week 108 (n=6) | -4.2 (10.87)
  Week 120 (n=1) | 4.2 (0)

42. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) General Health Perceptions Category: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=26) | 0.7 (14.27)
  Week 24 (n=25) | 3.8 (14.98)
  Week 36 (n=22) | 6.2 (15.99)
  Week 48 (n=19) | 7.2 (13.36)
  Week 60 (n=18) | 0.7 (10.65)
  Week 72 (n=15) | 9.1 (10.1)
  Week 84 (n=15) | 7.2 (13.03)
  Week 96 (n=11) | 10.9 (16)
  Week 108 (n=7) | 9 (16.61)
  Week 120 (n=3) | 4.7 (12.92)

43. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Change in Health Category: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=30) | 1.4 (1.75)
  Week 24 (n=29) | 1.7 (1.67)
  Week 36 (n=25) | 1.7 (1.8)
  Week 48 (n=22) | 1.7 (2.4)
  Week 60 (n=20) | 1.3 (2.57)
  Week 72 (n=16) | 1.6 (2.13)
  Week 84(n=16) | 1.3 (1.98)
  Week 96 (n=12) | 1.5 (2.02)
  Week 108 (n=8) | 0.9 (2.7)
  Week 120 (n=3) | 2.3 (0.58)

44. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Parental Impact - Emotional Category: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=30) | 11.4 (26.12)
  Week 24 (n=28) | 19 (28.59)
  Week 36 (n=26) | 29.2 (33.1)
  Week 48 (n=23) | 34.1 (33.98)
  Week 60 (n=20) | 31.7 (32.4)
  Week 72 (n=16) | 34.4 (36.37)
  Week 84 (n=16) | 27.6 (41.69)
  Week 96 (n=11) | 43.9 (40.15)
  Week 108 (n=8) | 46.9 (40.81)
  Week 120 (n=2) | 62.5 (41.25)

45. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Parental Impact - Time Category: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=30) | 4.6 (24.5)
  Week 24 (n=28) | 13.5 (28.59)
  Week 36 (n=26) | 21.8 (24.24)
  Week 48 (n=23) | 18.4 (24.76)
  Week 60 (n=20) | 13.3 (31.55)
  Week 72 (n=16) | 22.2 (30.09)
  Week 84 (n=16) | 17.4 (35.13)
  Week 96 (n=12) | 20.4 (27.15)
  Week 108 (n=8) | 15.3 (25.85)
  Week 120 (n=2) | 55.6 (62.85)

46. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Family Activities Category: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=30) | 8.3 (28.41)
  Week 24 (n=28) | 17.6 (24.15)
  Week 36 (n=26) | 20 (28.5)
  Week 48 (n=23) | 16.8 (26.43)
  Week 60 (n=20) | 14.8 (30.9)
  Week 72 (n=16) | 17.2 (31.43)
  Week 84 (n=16) | 18.2 (30.27)
  Week 96 (n=12) | 19.4 (27.6)
  Week 108 (n=8) | 20.8 (29.38)
  Week 120 (n=2) | 68.8 (20.62)

47. Secondary Outcome: Child's Health Questionnaire Parent Form (CHQ-PF50) Family Cohesion Category: Mean Change From Baseline to Each Visit
Description: as for outcome 33
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 32
units on a scale
  Week 12 (n=30) | 2.5 (14)
  Week 24 (n=28) | 4.3 (23.28)
  Week 36 (n=26) | 5.6 (20.66)
  Week 48 (n=23) | 3.7 (15.61)
  Week 60 (n=20) | 4.8 (16.66)
  Week 72 (n=16) | 7.2 (29.15)
  Week 84 (n=16) | 8.4 (39.19)
  Week 96 (n=12) | 18.8 (35.36)
  Week 108 (n=8) | 19.4 (35.3)
  Week 120 (n=2) | -27.5 (38.89)

ADVERSE EVENTS:
Time Frame: TEAEs were collected from first dose of study drug until 70 days after the last dose of study drug and before start of commercial adalimumab or other biologics (32.5 months); SAEs were collected from the time informed consent was obtained (33.5 months).
Description: A treatment-emergent AE (TEAE) is defined as any AE with onset or worsening reported by a participant from the time that the first dose of adalimumab is administered until 5 half-lives (70 days) have elapsed following discontinuation of adalimumab administration. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 5/32
Other Adverse Events (participants affected / at risk) | 27/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=32)
Dental caries (Gastrointestinal disorders) | 1
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1
Gastroenteritis rotavirus (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=32)
Arthropod bite (Injury, poisoning and procedural complications) | 2
Body temperature increased (Investigations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6
Headache (Nervous system disorders) | 2
Uveitis (Eye disorders) | 2
Pyrexia (General disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 4
Acute tonsillitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 6
Cystitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 4
Gastroenteritis viral (Infections and infestations) | 2
H1N1 influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 8
Otitis media (Infections and infestations) | 5
Pharyngitis (Infections and infestations) | 3
Pharyngitis streptococcal (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.